CLINICAL TRIAL: NCT04941638
Title: Comparison of Distal Radial, Proximal Radial and Femoral Access in ST-Segment Elevation Myocardial Infarction
Brief Title: Comparison of Vascular Access in STEMI
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yongcheol Kim, Professor, Yonsei University
Other Study IDs: DRA-STEMI
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-06

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Distal radial access; Snuffbox approach; ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Distal radial access — Vascular access for primary PCI in patients with STEMI
  Other Names: Proximal radial access; Femoral access

SUMMARY:
Distal radial access (DRA) has recently introduced and previous studies have demonstrated that it is feasible option, showing several advantages including less bleeding and access-site complications over proximal radial access (PRA). Previous study reported the feasibility of DRA as an alternative option for primary percutaneous coronary intervention (PCI) in STEMI patients without major complication. However, comparison study of each vascular access for primary PCI have not been conducted until now. Here, The investigators aim to compare the DRA, PRA and femoral access (FA), in terms of feasibility and safety, in patients with STEMI.

This is a retrospective study with patients who underwent primary PCI for STEMI between March 2020 to May 2021. The primary outcome of this study is the access-site complication including major bleeding requiring transfusion or surgery, hematoma and arterial occlusion.

DETAILED DESCRIPTION:
Recently, DRA has gained the interest of interventional cardiologists and previous studies have demonstrated several advantages including patient and operator comfort, shorter hemostasis duration, less bleeding, and access-site complications over PRA. More recently, randomized trial demonstrated that DRA prevents radial artery occlusion after the procedure compared with PRA. From this perspective, DRA could be considered an alternative access route for primary PCI in selected STEMI patients using potent P2Y12 inhibitors such as ticagrelor or prasugrel, or glycoprotein IIb/IIIa inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Between March 2020 to May 2021, patients who underwent primary PCI for STEMI at the Yongin Severance Hospital

Exclusion Criteria:

* Refractory cardiogenic shock requiring extracorporeal membrane oxygenation (ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent primary PCI for STEMI without ECMO
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
access-site complication | 1 month
  puncture site related complication

SECONDARY OUTCOMES:
The success rate of the puncture | Through procedure
  The success rate (%) of vascular puncture
The success rate of the primary PCI | Through procedure
  Success rate (%) = Successful primary PCI / All PCI procedures
The percentage of puncture time in Door-to-wiring time (%) | Through procedure
  Puncture time = time interval from local anesthesia induction to successful sheath cannulation.
  Door-to-wiring time = time elapsed from arrival of patient at the emergency department to guide wire passage through the lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Yongcheol Kim, Principal Investigator — Yongin Severance Hopistal
Locations (1):
- Yongin Severance Hospital, Yongin, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided